CLINICAL TRIAL: NCT04134975
Title: Evaluation of the Contribution of Intraoperative Scans Coupled With the Navigation for the Precision of the Positioning of the Pedicle Screws During a Lumbar Spine Surgery: a Prospective Randomised Study ScanRach Study
Brief Title: Evaluation of the Contribution of Intraoperative Scans Coupled With the Navigation for the Precision of the Positioning of the Pedicle Screws During a Lumbar Spine Surgery: a Prospective Randomised Study
Acronym: SCANRACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A01727-48
Record Dates: First submitted 2019-10-04; First posted 2019-10-22 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Lumbar Disc Disease; Surgical Procedure, Unspecified
Keywords: spin surgery; lumbar surgery; image guided surgery; radiation exposure; intraoperative navigation
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scanner Group (Experimental): lumbar spine surgical procedure with guided pedicle screw placement coupled with intraoperative scanning (BODYTOM, Samsung).
  Interventions: Procedure: Spine surgery
- fluoroscopy group (Active Comparator): lumbar spinal surgery with pedicle screw placement guided by fluoroscopy, a fluoroscopic control being performed with each set screw.
  Interventions: Procedure: Spine surgery

INTERVENTIONS:
Procedure: Spine surgery — surgery with pedicle screw placement between L1 and S1

SUMMARY:
Investigators team propose to evaluate the impact of the use of intraoperative scanning coupled with Stryker navigation, compared to the conventional fluoroscopy technique, on the accuracy of pedicle screws, in instrumented spinal surgery, by a randomised prospective study, in terms of pedicular screw accuracy. We will also evaluate the radiation exposure of the neurosurgical team and the patient in these two techniques.

DETAILED DESCRIPTION:
The use of pedicle screws in spinal surgery has seen a major advance in recent decades, allowing for greater biomechanical stability and higher fusion rates. In order to avoid any malposition that could cause neurological, vascular and visceral injuries and compromise this mechanical stability, imaging-guided surgical techniques have been developed. These are aimed at improving the positioning accuracy of pedicle screws to reduce these risks and improve mechanical stability and intervertebral fusion. Fluoroscopic examinations had long been the mainstay of intraoperative control imaging until the development of computer-assisted techniques. However, despite intraoperative examination, pedicle screw misalignment remains very common and even experienced surgeons can deviate screws in 5 to 20% of cases when using a standard fluoroscopic examination image. Thus, navigation techniques coupled with an intraoperative scanner, involving the acquisition of 2D images of the surgical field, have been developed. These techniques allow the neurosurgeon to navigate the spine and thus allow an improvement in the positioning accuracy of the pedicle screws. The correlate is an improvement of the safety of the procedure (reduction of complications) but also an optimisation of the biomechanical efficiency of the osteosynthesis.

With respect to the radiation emitted during navigated spinal surgery coupled with an intraoperative scan, some comparative studies have shown that the radiation rates received by the neurosurgical team and the patient were lower than the radiation rates received in conventional surgery. To date, few studies combining the analysis of the pedicular screw accuracy rate and the radiation rate transmitted to the neurosurgical team and patients have been published.

Therefore the team propose to evaluate the impact of the use of intraoperative scanning (BODYTom, Samsung) coupled with Stryker navigation, compared to the conventional fluoroscopy technique, on the accuracy of pedicle screws, in instrumented spinal surgery, by a randomised prospective study, in terms of pedicular screw accuracy. The investigator team will also evaluate the radiation exposure of the neurosurgical team and the patient in these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject over the age of 18
* Subject with lumbar degenerative pathology, requiring surgery with pedicle screw placement between L1 and S1, confirmed on MRI or preoperative scan
* Well conducted medical treatment, at least 3 months, which did not allow pain sedation
* Unprotected adult within the meaning of the law
* Subject belonging to a health insurance scheme
* Subject having signed their written informed consent.

Exclusion Criteria:

* Subject who is a minor, pregnant, parturient or breastfeeding woman
* Adult subject under legal protection, guardianship or deprivation of liberty by judicial or administrative decision
* Subject hospitalised without consent
* Medical contraindications to surgery and anaesthesia
* Contraindication of a medical nature to an MRI (pace-maker) or a scan being carried out
* Subject already treated by surgery for the same vertebral levels or adjacent levels
* Subject with scoliosis with a Cobb angle of more than 10°.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
pedicle screw positioning | 48 hours
  The accuracy of pedicle screw positioning will be evaluated on the early postoperative examination scan (within 48 hours after the intervention) and graded according to the following classification:
  * correctly positioned: pedicle screws perfectly positioned in the pedicle or with a deflection of less than 4mm.
  * poorly positioned: pedicle screws with a deflection greater than 4 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Private Hospital, Marseille, Paca, France